CLINICAL TRIAL: NCT04471584
Title: Comparative Analysis in Detection of Atrial Arrhythmia and Electrogram Quality in Three Different Insertable Cardiac Monitors
Brief Title: Comparative Analysis in Detection of Atrial Arrhythmia and ECG Quality in Three Different Insertable Cardiac Monitors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kansas City Heart Rhythm Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: KCHRF-ILR-0003
Record Dates: First submitted 2020-07-10; First posted 2020-07-15 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Arrhythmias, Cardiac
Keywords: Cardiac Arrhythmias; Implantable loop recorder; Comparative Analysis
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Abbott Confirm Rx (Active Comparator): All patients randomized to this group will be implanted Abbott Confirm RX
  Interventions: Device: Insertion of ILR device
- Medtronic Reveal LINQ (Active Comparator): All patients randomized to this group will be implanted Medtronic Reveal LINQ
  Interventions: Device: Insertion of ILR device
- Biotronik Biomonitor (Active Comparator): All patients randomized to this group will be implanted Biotronik Biomonitor
  Interventions: Device: Insertion of ILR device

INTERVENTIONS:
Device: Insertion of ILR device — All patients enrolled will be randomized to have one of three ILR devices implanted (BIOMONITOR III, Reveal LinQ, or Confirm RX) and will be given event monitoring device for concurrent evaluation.

SUMMARY:
Comparative analysis of available ILR devices models Abbot Confirm RxTM, Medtronic Reveal LINQTM, and Biotronik BIOMONITOR., evaluating detection performance and effective of transmission of these devices to better understand the differences between them.

DETAILED DESCRIPTION:
All devices have different algorithms for arrhythmia detection and structural design. Consequently, these devices vary in sensitivity of arrhythmia detection and data transmission.Therefore, we aim to expand a comparative analysis of available devices, evaluating detection performance and effective of transmission of these devices to better understand the differences between them.

ELIGIBILITY:
Inclusion Criteria:

Patients > 18 years of age with appropriate indication for ILR for atrial arrhythmia management.

Exclusion Criteria:

Inability to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Positive predictive values of device detected atrial arrhythmias | 12 months
  Positive predictive values of device detected atrial arrhythmias

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, Principal Investigator — Kansas City Heart Rhythm Research Foundation
Locations (1):
- Kansas City Heart Rhythm Institute, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parry SW, Matthews IG. Implantable loop recorders in the investigation of unexplained syncope: a state of the art review. Heart. 2010 Oct;96(20):1611-6. doi: 10.1136/hrt.2010.193417. PMID 20937748
- [Background] Palmisano P, Accogli M, Zaccaria M, Luzzi G, Nacci F, Anaclerio M, Favale S. Predictive factors for pacemaker implantation in patients receiving an implantable loop recorder for syncope remained unexplained after an extensive cardiac and neurological workup. Int J Cardiol. 2013 Oct 9;168(4):3450-7. doi: 10.1016/j.ijcard.2013.04.179. Epub 2013 May 20. PMID 23701932
- [Background] Pecha S, Aydin MA, Ahmadzade T, Hartel F, Hoffmann B, Steven D, Willems S, Reichenspurner H, Wagner FM. Implantable loop recorder monitoring after concomitant surgical ablation for atrial fibrillation (AF): insights from more than 200 continuously monitored patients. Heart Vessels. 2016 Aug;31(8):1347-53. doi: 10.1007/s00380-015-0735-4. Epub 2015 Aug 29. PMID 26319443
- [Background] Kapa S, Epstein AE, Callans DJ, Garcia FC, Lin D, Bala R, Riley MP, Hutchinson MD, Gerstenfeld EP, Tzou W, Marchlinski FE, Frankel DS, Cooper JM, Supple G, Deo R, Verdino RJ, Patel VV, Dixit S. Assessing arrhythmia burden after catheter ablation of atrial fibrillation using an implantable loop recorder: the ABACUS study. J Cardiovasc Electrophysiol. 2013 Aug;24(8):875-81. doi: 10.1111/jce.12141. Epub 2013 Apr 11. PMID 23577826
- [Background] Lauschke J, Busch M, Haverkamp W, Bulava A, Schneider R, Andresen D, Nagele H, Israel C, Hindricks G, Bansch D. New implantable cardiac monitor with three-lead ECG and active noise detection. Herz. 2017 Sep;42(6):585-592. doi: 10.1007/s00059-016-4492-7. Epub 2016 Oct 28. PMID 27796409
- [Background] Nolker G, Mayer J, Boldt LH, Seidl K, VAN Driel V, Massa T, Kollum M, Brachmann J, Deneke T, Hindricks G, Jung W, Brunner KJ, Kraus S, Hummer A, Lewalter T. Performance of an Implantable Cardiac Monitor to Detect Atrial Fibrillation: Results of the DETECT AF Study. J Cardiovasc Electrophysiol. 2016 Dec;27(12):1403-1410. doi: 10.1111/jce.13089. Epub 2016 Oct 7. PMID 27565119
- [Background] Ciconte G, Saviano M, Giannelli L, Calovic Z, Baldi M, Ciaccio C, Cuko A, Vitale R, Giacopelli D, Conti M, Lipartiti F, Giordano F, Maresca F, Moscatiello M, Vicedomini G, Santinelli V, Pappone C. Atrial fibrillation detection using a novel three-vector cardiac implantable monitor: the atrial fibrillation detect study. Europace. 2017 Jul 1;19(7):1101-1108. doi: 10.1093/europace/euw181. PMID 27702865
- [Background] Hindricks G, Pokushalov E, Urban L, Taborsky M, Kuck KH, Lebedev D, Rieger G, Purerfellner H; XPECT Trial Investigators. Performance of a new leadless implantable cardiac monitor in detecting and quantifying atrial fibrillation: Results of the XPECT trial. Circ Arrhythm Electrophysiol. 2010 Apr;3(2):141-7. doi: 10.1161/CIRCEP.109.877852. Epub 2010 Feb 16. PMID 20160169
- [Background] Lee R, Mittal S. Utility and limitations of long-term monitoring of atrial fibrillation using an implantable loop recorder. Heart Rhythm. 2018 Feb;15(2):287-295. doi: 10.1016/j.hrthm.2017.09.009. Epub 2017 Sep 13. PMID 28919290